CLINICAL TRIAL: NCT07281573
Title: The Effect of Exercises on the Shear Wave Velocity of the Median Nerve and the 3rd FDS in Patients With Carpal Tunnel Syndrome
Brief Title: Effect of Exercise on Ultrasound SWV in CTS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jošt Peterca, asst. Jošt Peterca MSc, researcher, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0120-25/2023/3
Record Dates: First submitted 2025-11-20; First posted 2025-12-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome; Peripheral Neuropathies
Keywords: CTS; Nerve gliding; strength; stiffness; Ultrasound; Shear wave velocity
MeSH Terms: conditions — Carpal Tunnel Syndrome; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: The investigators conducted a prospective, randomized, three-arm, parallel-group trial with a 1:1:1 allocation ratio to Gliding, Strength, and Control groups. Outcome measures were assessed before and after the intervention. Randomization of participants into two intervention groups and one control group was performed using the Clinical Trial Randomization Tool developed by the National Cancer Institute. The same tool was applied in participants with bilateral CTS to randomly determine which hand was assessed and included in the study.
Who Masked: Investigator
Masking Description: Ultrasound SWV measurements were performed by the primary investigator, who was blinded to participants' CTS diagnoses. A second investigator conducted the randomization process and scheduled participants' appointments; consequently, the primary investigator remained unaware of participant details prior to the SWV assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gliding group (Experimental): Participants randomized to Gliding received written description of exercises supported with images. Nerve and tendon gliding exercises targeted flexion and extension of the index and ring fingers, complemented by wrist flexion and extension movements. These exercises were taken from literature and designed to promote median nerve and tendon gliding through the carpal tunnel, thereby reducing entrapment of the median nerve and the third flexor digitorum superficialis (FDS) tendon (Abdolrazaghi et al., 2023; Savage & Albano, 2020; Sheereen et al., 2022).
  Interventions: Other: Nerve and tendon gliding exercises and strength exercises
- Strength group (Experimental): Patients randomized to Strength group received written description of exercises supported with images. Strengthening exercises involved movement patterns (finger and wrist flexion and extension) similar to the nerve and tendon gliding exercises; however, external resistance was introduced through the use of hand therapy resistance balls (Unver & Akyolcu, 2018) or low-weight dumbbells ranging from 0.5 to 2.0 kg depending on the participant (Doyle, 2024; Hamzeh et al., 2021).
  Interventions: Other: Nerve and tendon gliding exercises and strength exercises
- Control (No Intervention): The control group did not participate in any training program and was instructed to continue with their usual daily and work-related activities.

INTERVENTIONS:
Other: Nerve and tendon gliding exercises and strength exercises — The intervention lasted for 3 weeks and was performed once daily. Each participant recieved a detailed exercise plan including sets and repetitions and exercise description in steps and images of body parts position at each step of the exercise. The first session was demonstrated and supervised by a kinesiologist with 8 years of experiences. Nerve and tendon gliding exercises included the movements of arms, hands palms and fingers that triggered the gliding of the median nerve and 3rd FDS tendon through the carpal tunnel. There were 5 exercises for nerve gliding and 5 exercises for tendon gliding in the exercise plan. Furthermore the strength group exercise plan also included 5 exercises that were focusing on fingers and palm flexion and extension with therapeutic ball and elastic bands and wrist flexion and extension using low weight dumbbells (<2.0kg).
  Arms: Gliding group; Strength group

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral neuropathy, and studies suggest exercises can be used for symptom management. Purpose: The study evaluated the impact of exercise protocols on the ultrasound shear wave velocity (SWV) of the median nerve and 3rd flexor digitorum superficialis (3rd FDS) in participants with mild to moderate CTS. Methods: Ninety-one CTS participants (79 females) were divided into control group, nerve and tendon gliding exercise group, and strength exercise group. The participants followed a three-week daily exercise plan. The SWV measurements were conducted using Canon Aplio i800 ultrasound and linear probe (LX18i5). Regions of interest were positioned within the nerve epineurium and hyperechogenic borders of the 3rd FDS tendon. The pre- and post-intervention SWV values were recorded. Results: In preliminary results on a smaller sample, trends indicated reduced SWV in both the median nerve and 3rd FDS in the nerve and tendon gliding group and reduced SWV in the median nerve in the strengthening group. No measurable change was observed in the 3rd FDS in strength group and in the control group. Conclusion: Trends suggest specific exercises may decrease stiffness in the median nerve and 3rd FDS in CTS participants.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the impact of exercise protocols on the US SWV of the median nerve and 3rd FDS in the carpal tunnel in participants with mild to moderate CTS. The investigators aim to establish US SWE as a potential method to monitor nerve and tendon SWE changes due to exercise intervention and consequently show the effect of different exercise interventions on mechanical changes within the carpal tunnel.

This study was conducted in accordance with the ethical principles of the Declaration of Helsinki and Good Clinical Practice guidelines. The study protocol adhered to the CONSORT guidelines for reporting randomized trials and received approval from the National Medical Ethics Committee of the Republic of Slovenia (protocol number 0120-25/2023/3). Written informed consent was obtained from all participants prior to enrolment. Participants with suspected CTS were prospectively recruited from April 2025 to October 2025 at a single tertiary referral centre: the Institute of Clinical Neurophysiology, University Medical Centre Ljubljana, Slovenia. The inclusion criteria were as follows: (1) age between 24 and 78 years; (2) affirmative responses to at least two of the following three questions: (a) tingling in at least two of the first four digits; (b) symptoms worsening at night or in the morning; (c) symptom relief with hand flicking (flick sign); and (3) electrodiagnostic (EDx) confirmation of mild to moderate median nerve entrapment neuropathy at the wrist. Exclusion criteria were: (1) previous wrist fracture or surgery; (2) polyneuropathy, motor neuron disease, cervical radiculopathy, or brachial plexopathy; (3) structural abnormalities within the carpal tunnel; and (4) tenosynovitis. The investigators conducted a prospective, randomized, three-arm, parallel-group trial with a 1:1:1 allocation ratio to Gliding, Strength, and Control groups. Outcome measures were assessed before and after the intervention. Randomization of participants into two intervention groups and one control group was performed using the Clinical Trial Randomization Tool developed by the National Cancer Institute. The same tool was applied in participants with bilateral CTS to randomly determine which hand was assessed and included in the study.

The intervention lasted for 3 weeks and was performed once daily. The control group did not participate in any training program and was instructed to continue with their usual daily and work-related activities. Ultrasound SWV measurements were performed by the primary investigator, who was blinded to participants' CTS diagnoses. A second investigator conducted the randomization process and scheduled participants' appointments; consequently, the primary investigator remained unaware of participant details prior to the SWV assessment.

Participants randomized to Gliding or Strength group received written description of exercises supported with images. Nerve and tendon gliding exercises targeted flexion and extension of the index and ring fingers, complemented by wrist flexion and extension movements. These exercises were taken from literature and designed to promote median nerve and tendon gliding through the carpal tunnel, thereby reducing entrapment of the median nerve and the 3rd FDS tendon.

Strengthening exercises involved movement patterns (finger and wrist flexion and extension) similar to the nerve and tendon gliding exercises; however, external resistance was introduced through the use of hand therapy resistance balls or low-weight dumbbells ranging from 0.5 to 2.0 kg depending on the participant.

A contact phone number was provided in case of any difficulties. The first session was demonstrated and supervised by a kinesiologist with 8 years of experiences. After 7 days, participants were contacted by phone to assess their progress and discuss the potential symptoms issues related with exercise plan. Participants were seated with their forearms supinated, wrist in neutral position and fingers relaxed. Measurements were performed by a researcher with 3 years of experiences with ultrasound elastography using US system Canon Aplio i800 (Canon Medical Systems Europe BV, Zoetermeer, The Netherlands) with a i18Lx5 linear probe. Cross-sectional area (CSA) of the median nerve at the carpal tunnel inlet and at the forearm was measured. Thereafter, SWV of the median nerve and 3rd FDS tendon at the wrist was measured with the probe oriented longitudinally. Generous amount of gel was used to assure minimal pressure. Circular ROI was used and positioned within the epineurium of the median nerve and hyperechoic borders of the 3rd FDS tendon. SWV measurements were acquired only when the motion stability index (M-STB Index) displayed five consecutive green stars, indicating low or absent motion interference and stable image acquisition. The minimal time interval between two consecutive measurements was 10 seconds. Three consecutive SWV measurements were performed and median value in m/s was used for further analysis.

A sample size estimation was conducted for this randomized controlled trial, which included two intervention groups and one control group. Continuous outcomes were planned to be analyzed using pairwise comparisons between each intervention group and the control group. A two-sided significance level of 0.025 was applied to account for multiple comparisons using the Bonferroni correction. Assuming a statistical power of 0.80, an expected mean difference of 1.0, and a standard deviation of 1.25, the required sample size was estimated to be 30.14 participants per group. The calculation was performed using G*Power 3.1 software (Heinrich Heine University, Düsseldorf, Germany), based on effect sizes reported in previous randomized trials investigating exercise interventions for carpal tunnel syndrome.

Statistical analyses were performed using SPSS 29.0 (IBM Corp, Armonk, NY). Shapiro Wilk test was used to determine the variables normality distribution. For normal distributed variables, pre and post intervention SWV data was compared using ANOVA with within-subjects effect and interaction time vs. intervention. For group comparison, the investigators compared individual pairs of data with Paired sample T-test. Non-normally distributed variables were analysed using non-parametric Wilcoxon test. All statistical tests were two-tailed, with a p-value < 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age between 24 and 78 years
* tingling in at least two of the first four digits;
* symptoms worsening at night or in the morning;
* symptom relief with hand flicking (flick sign);
* electrodiagnostic (EDx) confirmation of mild to moderate median nerve entrapment neuropathy at the wrist.

Exclusion Criteria:

* previous wrist fracture or surgery;
* polyneuropathy,
* motor neuron disease,
* cervical radiculopathy,
* brachial plexopathy
* structural abnormalities within the carpal tunnel
* tenosynovitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Ultrasound shear wave velocity | SWV will be measured pre and post intervention in all three groups. There will be 3 weeks between pre and post intervention ultrasound SWV measurement
  SWV in m/s will be measured using ultrasound and linear probe i18Lx3. Three consequtive readings will be saved and the median value will be further procesed in statystical analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared to the repository of the University of Ljubljana at the stage of publication of the acquired data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD will be shared to the repository of the University of Ljubljana when the acquired IPD will be published in a scientific article
Access Criteria: Sign in to the repository with research ccredentials and account

REFERENCES:
- [Background] Wang Y, Qiang B, Zhang X, Greenleaf JF, An KN, Amadio PC, Zhao C. A non-invasive technique for estimating carpal tunnel pressure by measuring shear wave speed in tendon: a feasibility study. J Biomech. 2012 Nov 15;45(16):2927-30. doi: 10.1016/j.jbiomech.2012.09.002. Epub 2012 Sep 29. PMID 23031416
- [Background] Kubo K, Zhou B, Cheng YS, Yang TH, Qiang B, An KN, Moran SL, Amadio PC, Zhang X, Zhao C. Ultrasound elastography for carpal tunnel pressure measurement: A cadaveric validation study. J Orthop Res. 2018 Jan;36(1):477-483. doi: 10.1002/jor.23658. Epub 2017 Aug 14. PMID 28731271
- [Background] Bortolotto C, Lungarotti L, Fiorina I, Zacchino M, Draghi F, Calliada F. Influence of subjects' characteristics and technical variables on muscle stiffness measured by shear wave elastosonography. J Ultrasound. 2017 Mar 1;20(2):139-146. doi: 10.1007/s40477-017-0242-9. eCollection 2017 Jun. PMID 28593004
- [Background] Hobson-Webb LD, Massey JM, Juel VC, Sanders DB. The ultrasonographic wrist-to-forearm median nerve area ratio in carpal tunnel syndrome. Clin Neurophysiol. 2008 Jun;119(6):1353-7. doi: 10.1016/j.clinph.2008.01.101. Epub 2008 Apr 1. PMID 18387336
- [Background] Hamzeh H, Madi M, Alghwiri AA, Hawamdeh Z. The long-term effect of neurodynamics vs exercise therapy on pain and function in people with carpal tunnel syndrome: A randomized parallel-group clinical trial. J Hand Ther. 2021 Oct-Dec;34(4):521-530. doi: 10.1016/j.jht.2020.07.005. Epub 2020 Jul 30. PMID 32893098
- [Background] Unver S, Akyolcu N. The Effect of Hand Exercise on Reducing the Symptoms in Hemodialysis Patients with Carpal Tunnel Syndrome. Asian J Neurosurg. 2018 Jan-Mar;13(1):31-36. doi: 10.4103/ajns.AJNS_343_16. PMID 29492117
- [Background] Sheereen FJ, Sarkar B, Sahay P, Shaphe MA, Alghadir AH, Iqbal A, Ali T, Ahmad F. Comparison of Two Manual Therapy Programs, including Tendon Gliding Exercises as a Common Adjunct, While Managing the Participants with Chronic Carpal Tunnel Syndrome. Pain Res Manag. 2022 Jun 8;2022:1975803. doi: 10.1155/2022/1975803. eCollection 2022. PMID 35719196
- [Background] Savage NJ, Albano J. Marrying Tendon and Nerve Gliding Exercises with Hydrodissection Following Injection for Carpal Tunnel Syndrome - A New Treatment Approach? J Orthop Case Rep. 2020 Dec;10(9):38-46. doi: 10.13107/jocr.2020.v10.i09.1896. PMID 34169015
- [Background] Abdolrazaghi HA, Khansari M, Mirshahi M, Ahmadi Pishkuhi M. Effectiveness of Tendon and Nerve Gliding Exercises in the Treatment of Patients With Mild Idiopathic Carpal Tunnel Syndrome: A Randomized Controlled Trial. Hand (N Y). 2023 Mar;18(2):222-229. doi: 10.1177/15589447211006857. Epub 2021 Apr 15. PMID 33855879

DOCUMENTS (1):
  • Informed Consent Form (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT07281573/ICF_000.pdf